CLINICAL TRIAL: NCT02944617
Title: Assessment of the Role of Bifidobacterium-Containing Food Supplement Activia™ and Bacteriomic Profiling and Other Biomarkers Associated With Vascular Endothelial Growth Factor Tyrosine Kinase Inhibitor (VEGF-TKI)-Induced Diarrhea in Patients With Metastatic Renal Cell Carcinoma (mRCC)
Brief Title: Probiotic Yogurt Supplement in Reducing Diarrhea in Patients With Metastatic Kidney Cancer Being Treated With Vascular Endothelial Growth Factor-Tyrosine Kinase Inhibitor
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: City of Hope Medical Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 16088; NCI-2016-01068 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 16088 (Other: City of Hope Medical Center)
Record Dates: First submitted 2016-07-27; First posted 2016-10-26 (Estimated); Results first posted 2023-04-19 (Actual); Last update posted 2024-02-23 (Actual); Status verified 2024-01

CONDITIONS: Diarrhea; Metastatic Renal Cell Carcinoma; Stage IV Renal Cell Cancer
MeSH Terms: conditions — Diarrhea; Carcinoma, Renal Cell

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Arm I (probiotic yogurt supplement) (Experimental): Patients receive probiotic supplement Activia yogurt QD during weeks 2-13 of VEGF-TKI treatment.
  Interventions: Other: Laboratory Biomarker Analysis; Dietary Supplement: Micronutrient-Fortified Probiotic Yogurt; Drug: VEGF-TKI
- Arm II (no intervention) (Active Comparator): Patients avoid any intake of yogurt or yogurt-containing foods and refrain from taking/consuming other probiotic supplements for 3 months.
  Interventions: Other: Laboratory Biomarker Analysis; Drug: VEGF-TKI

INTERVENTIONS:
Other: Laboratory Biomarker Analysis — Correlative studies
Dietary Supplement: Micronutrient-Fortified Probiotic Yogurt — Receive Activia yogurt
  Arms: Arm I (probiotic yogurt supplement)
Drug: VEGF-TKI — Must be received as standard of care chemotherapy

SUMMARY:
This randomized clinical trial studies how well probiotic yogurt supplement works in reducing diarrhea in patients with kidney cancer that has spread from the primary site to other places in the body (metastatic) and that are being treated with vascular endothelial growth factor-tyrosine kinase inhibitor therapy. Studying samples of blood and stool from patients who eat probiotic yogurt and those who avoid probiotic yogurt may help doctors plan better treatment.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To determine if adding Activia yogurt (containing Bifidobacterium lactis DN-173 010) to the diet of patients with metastatic renal cell carcinoma (mRCC) increases the level of Bifidobacterium spp in stool.

SECONDARY OBJECTIVES:

I. To determine if Activia reduces the incidence of diarrhea for mRCC patients treated with vascular endothelial growth factor - tyrosine kinase inhibitor (VEGF-TKI) therapy.

II. To compare pre-treatment levels of circulating T regulatory (Treg) cells and levels of peripheral signal transducers and activators of transcription 3 (STAT3) in patients with and without diarrhea with VEGF-TKI therapy, and correlate with Bifidobacterium, other bacteria, and Activia.

III. To determine if patients with the diarrhea in mRCC patients treated with VEGF-TKI therapy have a lower baseline of Bifidobacterium spp.

IV. To assess the change in global stool bacteriomic profile of patients receiving therapy with VEGF-TKI therapy with or without Activia.

V. To better assess the feasibility of stool collection and bacteriomic profiling.

VI. To explore association between psychosocial symptoms (anxiety and depression) and bacteriomic profile and gastrointestinal toxicity in mRCC patients receiving VEGF-TKI therapy therapy.

OUTLINE: Patients are randomized to 1 of 2 arms.

ARM I: Patients receive probiotic supplement Activia yogurt twice daily (QD) during weeks 2-13 of VEGF-TKI treatment.

ARM II: Patients avoid any intake of yogurt or yogurt-containing foods and refrain from taking/consuming other probiotic supplements for 3 months.

ELIGIBILITY:
Inclusion Criteria:

* Cytologically or pathologically verified diagnosis of renal cell carcinoma (RCC)
* Diagnosis of RCC that is defined as metastatic by standard criteria (American Joint Committee on Cancer [AJCC] 7th edition, 2010)
* Planned treatment with any VEGF-TKI, treatment has not yet begun
* Ability to understand and the willingness to sign a written informed consent
* Ability to read and write English
* Documented consent to participation to include the following study specific procedures:

  * Be able to provide up to six serial stool collections at home and deliver to FedEx location that day as per standard operating procedure
  * Have three 10-ml blood samples taken during a routine clinic visit
  * To not take probiotic supplements except as oriented
  * If randomized to the probiotic-supplemented group (the yogurt-based supplement Activia), be willing to comply with daily intake and record this intake as a component of a dietary log; the patient will be asked not to take any yogurt or yogurt-containing foods beyond this
  * If randomized to the probiotic-restricted group, agree not to consume yogurt or yogurt-containing foods
  * Maintain a dietary log and stool frequency log

Exclusion Criteria:

* Patients with a known intolerance to lactose or other constituents of Activia
* Patients with irritable bowel syndrome, Crohn's disease, or other clinically significant gastrointestinal (GI) related condition that might confound the VEGF-TKI-related-diarrhea endpoint
* Patients taking antibiotics or who plan to begin taking antibiotics
* Any other condition that would, in the investigator's judgment, contraindicate the patient's participation in the clinical study due to safety concerns or compliance with clinical study procedures (including compliance issues related to feasibility/logistics)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2016-11-11 (Actual); Primary Completion 2021-12-19 (Actual); Study Completion 2021-12-19 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sumanta Pal, Principal Investigator — City of Hope Medical Center
Locations (1):
- City of Hope Medical Center, Duarte, California, United States

REFERENCES:
- [Derived] Dizman N, Hsu J, Bergerot PG, Gillece JD, Folkerts M, Reining L, Trent J, Highlander SK, Pal SK. Randomized trial assessing impact of probiotic supplementation on gut microbiome and clinical outcome from targeted therapy in metastatic renal cell carcinoma. Cancer Med. 2021 Jan;10(1):79-86. doi: 10.1002/cam4.3569. Epub 2020 Nov 1. PMID 33135866

RESULTS

PARTICIPANT FLOW:
Groups:
- Arm I (Probiotic Yogurt Supplement): Patients receive 4 oz. probiotic supplement Activia yogurt bid during weeks 2-13 and refrain from taking/consuming other probiotic supplements.
  Micronutrient-Fortified Probiotic Yogurt: Receive Activia yogurt
  VEGF-TKI: Must be received as standard of care chemotherapy
Period: Overall Study
Arm/Group | Arm I (Probiotic Yogurt Supplement) | Arm II (no Intervention)
Started | 11 | 10
Completed | 10 | 10
Not Completed | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Arm I (Probiotic Yogurt Supplement) | Arm II (no Intervention) | Total
Number analyzed (Participants) | 10 | 10 | 20
Age, Continuous [Median (Full Range); unit: years] | 67.0 [57 to 81] | 67.5 [32 to 78] | 67.5 [32 to 81]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 3 | 5
  Male | 8 | 7 | 15
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United States | 10 | 10 | 20

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Overall Response
Description: Per Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.1) for target lesions and assessed by MRI: Complete Response (CR), Disappearance of all target lesions; Partial Response (PR), >=30% decrease in the sum of the longest diameter of target lesions; Overall Response (OR) = CR + PR
Time Frame: Up to 3 years
Measure: Count of Participants; unit: Participants
Arm/Group | Arm I (Probiotic Yogurt Supplement) | Arm II (no Intervention)
Number analyzed (Participants) | 10 | 10
Participants | 2 | 1

2. Primary Outcome: Number of Participants With Diarrhea
Description: The rate of all grade diarrhea as graded by the Common Terminology Criteria for Adverse Events version 4.0 will be compared in the patients who receive the dietary supplement and those who do not. A Fisher's exact test with a 0.050 one-sided significance level will be used.
Time Frame: Up to 13 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Arm I (Probiotic Yogurt Supplement) | Arm II (no Intervention)
Number analyzed (Participants) | 10 | 10
Participants | 4 | 4
Statistical Analysis 1: Comparison: Arm I (Probiotic Yogurt Supplement) vs Arm II (no Intervention); Test type: Other; p = 1.00, Fisher Exact

3. Secondary Outcome: Clinical Benefit Rate
Description: Per Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.1) for target lesions and assessed by MRI:
  Complete Response (CR), Disappearance of all target lesions; Partial response (PR): At least a 30% decrease in the sum of diameters of all target lesions, taking as reference the baseline sum of diameters, in the absence of CR; Stable disease (SD): Neither sufficient shrinkage to qualify for CR or PR nor sufficient increase to qualify for PD; Progressive disease (PD): At least a 20% increase in the sum of diameters of target lesions, taking as reference the smallest sum of diameters on study (including baseline). Clinical Benefit Rate (CBR) = CR + PR + SD at 6 months
Time Frame: Up to 6 months
Measure: Number; unit: percentage of participants
Arm/Group | Arm I (Probiotic Yogurt Supplement) | Arm II (no Intervention)
Number analyzed (Participants) | 10 | 10
percentage of participants | 70 | 80

4. Secondary Outcome: Progression-free Survival (PFS)
Description: Estimated using the product-limit method of Kaplan and Meier. Failure defined as disease progression or death from any cause. Progression is defined using Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.1), as a 20% increase in the sum of the longest diameter of target lesions, or a measurable increase in a non-target lesion, or the appearance of new lesions.
Time Frame: Up to 36 months
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Arm I (Probiotic Yogurt Supplement) | Arm II (no Intervention)
Number analyzed (Participants) | 10 | 10
Months | 6.2 [2.2 to 10.3] | 13.8 [6.2 to 21.5]
Statistical Analysis 1: Comparison: Arm I (Probiotic Yogurt Supplement) vs Arm II (no Intervention); Test type: Other; p = 0.077, Log Rank

ADVERSE EVENTS:
Time Frame: Adverse events were assessed from the time of initial treatment until 30 days post discontinuation of treatment, up to 4 months.
Arm/Group | Arm I (Probiotic Yogurt Supplement) | Arm II (no Intervention)
All-Cause Mortality (participants affected / at risk) | 3/10 | 6/10
Serious Adverse Events (participants affected / at risk) | 0/10 | 0/10
Other Adverse Events (participants affected / at risk) | 9/10 | 8/10
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm I (Probiotic Yogurt Supplement) (N=10) | Arm II (no Intervention) (N=10)
Transaminitis (Investigations) | 1 (1) | 0 (0)
Hypertension (General disorders) | 0 (0) | 2 (2)
Hand-foot Syndrome (Immune system disorders) | 1 (1) | 2 (2)
Sinusitis (General disorders) | 0 (0) | 1 (1)
Mucositis (General disorders) | 1 (1) | 2 (2)
Hypothyroidism (Endocrine disorders) | 0 (0) | 1 (1)
Fatigue (General disorders) | 1 (1) | 0 (0)
Gastritis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Colitis (Gastrointestinal disorders) | 1 (1) | 2 (2)
Epistaxis (General disorders) | 0 (0) | 1 (1)
Dermatitis (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Constipation (Gastrointestinal disorders) | 1 (1) | 0 (0)
Diarhea (Gastrointestinal disorders) | 4 (4) | 4 (4)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-06-12): https://cdn.clinicaltrials.gov/large-docs/17/NCT02944617/Prot_SAP_000.pdf